CLINICAL TRIAL: NCT06615661
Title: An Observational Real-World Evidence Study of Ab-Interno Goniotomy Performed Using the C-Rex Instrument in Patients With Primary Open Angle Glaucoma
Brief Title: A Real-World Evidence Study of Goniotomy With the C-REX™ Instrument in Patients With Primary Open Angle Glaucoma
Acronym: CIRCLE
Status: Recruiting | Type: Observational
Sponsor: Iantrek, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ITR-GON-041
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: Ocular Hypertension; Eye Diseases; Glaucoma; Goniotomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Eye Diseases; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- C-Rex surgery - combination: C-Rex surgery combined with cataract extraction/intraocular lens (IOL) implantation
  Interventions: Device: C-Rex Instrument
- C-Rex surgery - standalone: C-Rex surgery as a standalone intervention
  Interventions: Device: C-Rex Instrument

INTERVENTIONS:
Device: C-Rex Instrument — The C-Rex Instrument is a manual ophthalmic surgical instrument used for ab interno goniotomy and inner wall trabeculotomy.

SUMMARY:
This study enrolls adults with primary open angle glaucoma (POAG) who underwent goniotomy intraocular pressure (IOP)-lowering surgery with the C-Rex Instrument. Patients are consented prior to surgery and followed for 12 months postoperatively. Data regarding IOP, use of glaucoma medications, and any device-related complications are collected during the study time period.

DETAILED DESCRIPTION:
This a multicenter, observational real-world evidence study of eligible adults with primary open angle glaucoma (POAG) in whom ab-interno goniotomy surgery with the C-Rex Instrument was performed.

Data is collected from the preoperative visit(s) that directly preceded the surgery, the surgical procedure, and post-surgical visits through 12 months postoperatively.

Specific data collected includes C-Rex Instrument goniotomy surgical details, preoperative and postoperative IOP and use of ocular hypotensive medications, and device-related safety events.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Goniotomy surgery performed using the C-Rex Instrument

Exclusion Criteria:

* History of intraocular surgery within 8 weeks prior to C-Rex surgery
* Preoperative IOP higher than 33 mmHg
* Presence of a glaucoma type other than POAG
* Presence of clinically significant intraocular pathology other than cataract or glaucoma

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants who underwent IOP-lowering surgical procedures using the C-Rex Instrument to perform ab-interno goniotomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percent of eyes with intraocular pressure (IOP)reduction ≥20%in comparison with baseline. | 12 month postoperative
  Intraocular pressure (IOP) is at least 20% lower than before surgery without additional ocular hypotensive medications or IOP-lowering surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Omni Eye Services, Atlanta, Georgia
  - CIRCLE Site 04, Crossville, Tennessee

IPD SHARING:
Plan to Share IPD: No